CLINICAL TRIAL: NCT01244594
Title: The Effects of Two Functional Electrical Stimulation Cycling Paradigms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: The Craig H. Neilsen Foundation (Other); Magee Rehabilitation Hospital (Unknown); Temple University (Other); University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 164600
Record Dates: First submitted 2010-11-15; First posted 2010-11-19 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Cycling; Functional Electrical Stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High cadence, low resistance (Experimental): Subjects in this arm will cycle with functional electrical stimulation at a higher cadence (speed) and a lower resistance.
  Interventions: Other: Cycling with functional electrical stimulation
- Low cadence, high resistance (Experimental): Subjects in this arm will cycle with functional electrical stimulation at a lower cadence (speed) and a higher resistance.
  Interventions: Other: Cycling with functional electrical stimulation

INTERVENTIONS:
Other: Cycling with functional electrical stimulation — Subjects will cycle with functional electrical stimulation for one hour, 3 times per week at Magee Rehab's outpatient center. Subjects will cycle for a total of 26 weeks (6 months).

SUMMARY:
Background:

People with spinal cord injury (SCI) are at risk for many health conditions, some of which can be decreased with exercise. Cycling with Functional Electrical Stimulation (FES) is one way to obtain exercise after SCI. However, cycling with FES has only been done one way, which involves pedaling more quickly with less force to work against. Pedaling more slowly would allow the person to work against more force, which may lead to greater improvements in bone mineral density and muscle size. It may also lead to greater changes in bone make-up, body fat, and cholesterol levels. All of these improvements may lead to a decrease in bone fractures and cardiovascular disease, two major medical issues that exist in the SCI population. Study Aims: This study will compare the outcomes on bone, muscle and cardiovascular health between the commonly used method of pedaling more quickly to a new method of pedaling more slowly. Both groups will work against the maximal force possible. It is expected that the group pedaling more slowly will work against greater force and thus will have improved outcomes compared to other group pedaling faster. Methods: Twenty people with SCI, ages 18-65 years, will be randomly assigned to a treatment group and will participate in three 60-minute sessions per week for 6 months at an outpatient rehabilitation center. All subjects must have complete paralysis of both legs, but may have sensation preserved. Before and after 6 months of exercise, subjects will have an MRI scan to assess muscle size and bone, a dexascan to assess bone, a strength test using electrical stimulation to assess muscle force, an analysis of fat free body tissue, and lab work to measure cholesterol, bone factors that provide insight into bone change, and nutritional status. Relevance: If the protocol of pedaling more slowly results in greater improvements, this technique can be applied to clinical practice. Some people with SCI have FES cycles in their homes and many have been cycling for many years. This new technique may allow them to obtain more benefits than what they currently are receiving from FES cycling. In addition, it is important to maintain overall bone, muscle and cardiovascular health so that people with SCI are health and ready when spinal cord regeneration becomes clinically available.

ELIGIBILITY:
Inclusion Criteria:

* Cervical or thoracic SCI of greater than 6 months duration
* American Spinal Injury Association Impairment Scale (AIS) levels A (motor and sensory complete) or B (motor complete)
* Intact lower motor neurons to the quadriceps, hamstrings, and gluteal muscles

Exclusion Criteria:

* History of renal or bladder stones or renal impairment
* Presence of conditions that require chronic steroids
* Symptomatic or known cardiac disease
* Pulmonary disease limiting exercise tolerance
* Ventilator dependency
* Implanted devices that may be adversely affected by the FES system
* Lower extremity fragility fractures in the previous 3 months
* Severe spasticity in legs
* Presence of a Grade 2 or higher pressure ulcer
* Severely limited range of joint motion
* Heterotopic ossification of joints in the lower extremities
* Uncontrolled autonomic dysreflexia
* Dislocation of one or both hips
* Pregnancy or plans to become pregnant during the study
* Post menopausal, if female
* Current seizure disorder
* Participation in activities involving electrical stimulation or activity based therapy within the past 3 months
* Participation in a neuroregenerative intervention within the past 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Bone density and bone microarchitecture | Baseline
  Bone is measured using dexascan and Magnetic Resonance Imaging (MRI) to examine different types of bone (cortical and trabecular).
Bone density and bone microarchitecture | 6 months
  Bone is measured using dexascan and Magnetic Resonance Imaging (MRI) to examine different types of bone (cortical and trabecular).
Muscle volume | Baseline
  Muscle volume is assessed using MRI
Muscle volume | 6 months
  Muscle volume is assessed using MRI

SECONDARY OUTCOMES:
Muscle strength | Baseline
  Muscle strength is assessed by stimulating the muscle using a max twitch technique and measuring the isometric force output on a dynamometer.
Muscle strength | 3 months
  Muscle strength is assessed by stimulating the muscle using a max twitch technique and measuring the isometric force output on a dynamometer.
Muscle strength | 6 months
  Muscle strength is assessed by stimulating the muscle using a max twitch technique and measuring the isometric force output on a dynamometer.
Bone markers | baseline
  Bone markers are assessed through blood and urine analysis.
Bone markers | 3 months
  Bone markers are assessed through blood and urine analysis.
Bone markers | 6 months
  Bone markers are assessed through blood and urine analysis.
Fat free soft tissue | baseline
  Fat free mass is assessed using a bioimpedance monitor.
Fat free soft tissue | 3 months
  Fat free mass is assessed using a bioimpedance monitor.
Fat free soft tissue | 6 months
  Fat free mass is assessed using a bioimpedance monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Therese E Johnston, PT, PhD, MBA, Principal Investigator — Thomas Jefferson University
Locations (3):
- United States (3):
  - Magee Rehabilitation Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Johnston TE, Marino RJ, Oleson CV, Schmidt-Read M, Leiby BE, Sendecki J, Singh H, Modlesky CM. Musculoskeletal Effects of 2 Functional Electrical Stimulation Cycling Paradigms Conducted at Different Cadences for People With Spinal Cord Injury: A Pilot Study. Arch Phys Med Rehabil. 2016 Sep;97(9):1413-1422. doi: 10.1016/j.apmr.2015.11.014. Epub 2015 Dec 17. PMID 26705884